CLINICAL TRIAL: NCT00818766
Title: Extended Antibiotic Prophylaxis for the Prevention of Infectious Complications Associated With Tube Thoracostomy in Patients Undergoing Elective General Thoracic Surgery: A Double-Blind, Placebo-Controlled, Randomized Trial
Brief Title: Efficacy of Post-operative Antibiotic Prophylaxis for Thoracic Surgery Requiring Tube Thoracostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, David A. Oxman, MD, Co-Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007p002164
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Results first posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-03

CONDITIONS: Antibiotic Prophylaxis
Keywords: Thoracic Surgery; Antibiotic Prophylaxis; Chest Tube
MeSH Terms: interventions — Cefazolin; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antibiotic (Active Comparator): Participants received intravenous (IV) cefazolin or vancomycin (for participants allergic to cephalosporin) immediately following surgery for 48 hours or until all chest tubes were removed, whichever occurred first.
  Interventions: Drug: cefazolin or vancomycin
- Placebo (Placebo Comparator): Participants received IV placebo-matching antibiotics immediately following surgery for 48 hours or until all chest tubes were removed, whichever occurred first.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: cefazolin or vancomycin — Cefazolin IV every eight hours post-operatively for 48 hours or until all chest tubes were removed, whichever occurred first. Participants under 80 kg received 1 gram of cefazolin and participants who were 80 kg or more received 2 grams of cefazolin. Participants who were penicillin-allergic received 1 gram of vancomycin every 12 hours for 48 hours or until all chest tubes were removed, whichever occurred first.
  Other Names: Cefazolin (Ancef); Vancomycin (Vancocin)
  Arms: Antibiotic
Drug: Placebo — Participants received IV placebo for 48 hours post-operatively or until all chest tubes were removed, whichever occurred first.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate if post-operative antibiotic prophylaxis decreases infectious complications when compared to pre-operative antibiotics alone, in patients undergoing elective thoracic surgery requiring tube thoracostomy (chest tube).

DETAILED DESCRIPTION:
There is currently no evidence-based standard for the extended use of prophylactic antibiotics in patients receiving thoracic surgery that results in the placement of a tube thoracostomy (chest tube). The rationale for this prophylaxis is that antibiotics directed at typical skin flora may reduce the rate of infectious complications, such as surgical site infection and empyema.

Currently, clinicians' approach to post-operative antibiotic prophylaxis in patients undergoing tube thoracostomy associated with thoracic and cardio-thoracic surgery varies widely. While reducing the infectious complications of thoracic surgery is an important goal, it is also important to reduce the use of unnecessary antibiotics. As there is equipoise on the benefit of extended antibiotic prophylaxis for tube thoracostomy, our study will examine two prevailing clinical practices and attempt to determine if one leads to better patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older undergoing elective thoracic surgery at Brigham & Women's Hospital. The majority of these patients will be undergoing lung resection for either the evaluation of a lung mass, or for the removal of a known malignancy. Some participants may be undergoing biopsy or removal of a mediastinal mass.
* Undergoing thoracic surgery procedure expected to require tube thoracostomy.
* Ability to give informed consent

Exclusion Criteria:

* Patients undergoing the following complex thoracic surgical procedures:

  * Pneumonectomy
  * Decortication
  * Chemical pleurodesis
  * Pleurectomy
  * Lung volume reduction
  * Esophagectomy
* Patients with the following conditions:

  * Prior diagnosis of empyema or lung abscess.
  * Cystic fibrosis
  * Known or suspected pneumonia pre-operatively.
  * Known hypersensitivity to beta-lactam antibiotics and vancomycin
  * Current or recent antibiotic use within one week of surgery.
  * Anticipated requirement for postoperative antibiotic in addition to 48 hours of cefazolin or vancomycin.
  * Renal insufficiency with estimated creatinine clearance <60 ml/minute.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2008-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Baden, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Oxman DA, Issa NC, Marty FM, Patel A, Panizales CZ, Johnson NN, Licona JH, McKenna SS, Frendl G, Mentzer SJ, Jaklitsch MT, Bueno R, Colson Y, Swanson SJ, Sugarbaker DJ, Baden LR. Postoperative antibacterial prophylaxis for the prevention of infectious complications associated with tube thoracostomy in patients undergoing elective general thoracic surgery: a double-blind, placebo-controlled, randomized trial. JAMA Surg. 2013 May;148(5):440-6. doi: 10.1001/jamasurg.2013.1372. PMID 23325435

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients presenting for elective lung surgery and expected to require tube thoracostomy were approached for participation in the study at the time of preoperative evaluation.
Groups:
- Antibiotic: Cefazolin or vancomycin: Cefazolin IV every eight hours post-operatively for 48 hours or until all chest tubes were removed, whichever occurred first. Participants under 80 kg received 1 gram of cefazolin and participants who were 80 kg or more received 2 grams of cefazolin. Participants who were cephalosporin-allergic received 1 gram of vancomycin every 12 hours for 48 hours or until all chest tubes were removed, whichever occurred first.
Period: Overall Study
Arm/Group | Antibiotic | Placebo
Started | 125 | 126
Received Allocated Intervention | 122 (1 withdrew consent, 1 had active infection and 1 was given open-label antibiotic after surgery.) | 126
Intent-to-Treat Population | 121 (1 participant was randomized twice but only counted once (per first randomization).) | 124 (2 participants were randomized twice but only counted once (per first randomization).)
Completed (Completed = completed through 28-day follow-up phone call) | 110 | 116
Not Completed | 15 | 10
Not completed — Could not be Contacted on Day 28 | 11 | 10
Not completed — Death | 1 | 0
Not completed — Did not Receive Allocated Intervention | 3 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) Population included all participants who were randomized and received their allocated intervention. 1 participant in the antibiotic arm and 2 participants in the placebo arm were randomized twice but are only counted once (per their first randomization) in the ITT Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Antibiotic | Placebo | Total
Number analyzed (Participants) | 121 | 124 | 245
Age, Continuous [Median (Full Range); unit: years] | 63 [24 to 85] | 62 [26 to 84] | 62.5 [24 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 70 | 139
  Male | 52 | 54 | 106

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced At Least One Postoperative Infectious Complication
Description: Infectious complications include: surgical site infection, empyema, pneumonia, and the occurrence of Clostridium difficile colitis within 28 days of surgery. Participants are only counted once regardless of how many different infectious complications they had.
Time Frame: Up to 28 days after surgery
Population: Intent-to-Treat (ITT) Population included all participants who were randomized and received their allocated intervention. 1 participant in the antibiotic arm and 2 participants in the placebo arm were randomized twice but are only counted once (per first randomization) in the ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotic | Placebo
Number analyzed (Participants) | 121 | 124
Participants | 13 | 8
Statistical Analysis 1: Comparison: Antibiotic vs Placebo; Test type: Superiority or Other; p = .26, Fisher Exact; Risk Difference (RD) = -4.3, 95% CI [-11.3 to 2.7]

2. Primary Outcome: Number of Participants Who Experienced Surgical Site Infection
Description: Surgical Site Infection:
  1. Superficial surgical site infection - involves only skin or subcutaneous tissue around incision and has at least one of the following criteria:
     * purulent drainage
     * organisms isolated from aseptically obtained culture
     * pain or tenderness, localized swelling, redness or heat and the incision deliberately opened by a surgeon
     * diagnosis of a superficial wound infection by a surgeon
  2. Deep surgical site infection - involves deep soft tissues e.g. fascia or muscle and has at least one of the following:
     * purulent drainage from the incision but not from the organ/space of the surgical site
     * deep incision spontaneously dehisces or deliberately opened by surgeon when patient has at least one of following signs or symptoms - fever (>38°C), localized pain or tenderness.
     * an abscess or evidence of infection involving incision is found on direct examination, histopathologic or radiographic examination
     * diagnosis of a deep wound infection
Time Frame: Up to 28 days after surgery
Population: ITT Population included all participants who were randomized and received their allocated intervention. 1 participant in the antibiotic arm and 2 participants in the placebo arm were randomized twice but are only counted once (per first randomization) in the ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotic | Placebo
Number analyzed (Participants) | 121 | 124
Participants | 6 | 5
Statistical Analysis 1: Comparison: Antibiotic vs Placebo; Test type: Superiority or Other; p = 0.77, Fisher Exact; Risk Difference (RD) = -0.93, 95% CI 2-sided [-6.1 to 4.3]

3. Primary Outcome: Number of Participants Who Experienced Pneumonia
Description: Pneumonia:
  A new infiltrate on chest x-ray associated with at least three of the following:
  * fever (>38°C)
  * purulent sputum
  * leukopenia (white blood cell [WBC] count of <4000/µL) or leukocytosis (WBC count of >11000/µL)
  * sputum culture with pathogenic bacteria
  * increased oxygen requirements
Time Frame: Up to 28 days after surgery
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotic | Placebo
Number analyzed (Participants) | 121 | 124
Participants | 7 | 3
Statistical Analysis 1: Comparison: Antibiotic vs Placebo; Test type: Superiority or Other; p = .21, Fisher Exact; Risk Difference (RD) = -3.4, 95% CI 2-sided [-8.3 to 1.6]

4. Primary Outcome: Number of Participants Who Experienced Empyema
Description: Empyema:
  Positive pleural culture result or purulence within the thoracic space and leukocytosis or fever (>38°C).
Time Frame: Up to 28 days after surgery
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotic | Placebo
Number analyzed (Participants) | 121 | 124
Participants | 1 | 0
Statistical Analysis 1: Comparison: Antibiotic vs Placebo; Test type: Superiority or Other; p = .49, Fisher Exact

5. Primary Outcome: Number of Participants Who Experienced Clostridium (C) Difficile Colitis
Description: C. Difficile Colitis:
  Positive for C difficile toxin assay results and any 1 of the following:
  * new diarrhea
  * ileus or toxic megacolon
  * leukopenia (WBC count of <4000/µL) or leukocytosis (WBC count of >11000/µL)
  * findings from sigmoidoscopy, colonoscopy, or histopathologic examination consistent with C difficile infection
Time Frame: Up to 28 days after surgery
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotic | Placebo
Number analyzed (Participants) | 121 | 124
Participants | 0 | 0

6. Secondary Outcome: Number of Participants Who Received Additional Antibiotics for Any Reason Within 28 Days After Surgery
Description: The number of participants who needed any additional non-study antibiotics for any reason after randomization.
Time Frame: Up to 28 days after surgery
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotic | Placebo
Number analyzed (Participants) | 121 | 124
Participants | 32 | 31
Statistical Analysis 1: Comparison: Antibiotic vs Placebo; Test type: Superiority or Other; p = .25, Fisher Exact

7. Secondary Outcome: Number of Participants Who Needed Reoperation
Description: The number of participants who needed reoperations for any reason from the time after the first surgery to the end of the 28-day follow-up period.
Time Frame: Up to 28 days after surgery
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotic | Placebo
Number analyzed (Participants) | 121 | 124
Participants | 5 | 10
Statistical Analysis 1: Comparison: Antibiotic vs Placebo; Test type: Superiority or Other; p = .25, Fisher Exact

8. Secondary Outcome: Length of Hospital Stay
Description: The length of hospital stay is the number of days the participant remained in the hospital.
Time Frame: From day of surgery to discharge (up to 35 days)
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | Antibiotic | Placebo
Number analyzed (Participants) | 121 | 124
days | 3 [1 to 35] | 3 [0 to 31]

9. Secondary Outcome: Time to Removal of Chest Tubes
Description: Time to removal of chest tubes is the number of days from the time of chest tube placement to time they were removed.
Time Frame: From day of surgery to removal of chest tubes (up to 33 days)
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | Antibiotic | Placebo
Number analyzed (Participants) | 121 | 124
days | 2 [0 to 32] | 2 [0 to 33]

10. Secondary Outcome: Number of Participants With Allergic Reactions
Description: The number of participants with an allergic reaction to a drug.
Time Frame: Up to 28 days after surgery
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotic | Placebo
Number analyzed (Participants) | 121 | 124
Participants | 0 | 0

11. Secondary Outcome: All-Cause Mortality
Description: All-cause mortality is the number of deaths that occurred during the study period, regardless of the cause.
Time Frame: Up to 28 days after surgery
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotic | Placebo
Number analyzed (Participants) | 121 | 124
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: From the time immediately following surgery up to 28 days.
Arm/Group | Antibiotic | Placebo
All-Cause Mortality (participants affected / at risk) | 1/121 | 0/124
Serious Adverse Events (participants affected / at risk) | 1/121 | 0/124
Other Adverse Events (participants affected / at risk) | 0/121 | 0/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antibiotic (N=121) | Placebo (N=124)
Atrial fibrillation (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No